CLINICAL TRIAL: NCT01035372
Title: Pilot Study on the Tolerability of Dietary Dried Plum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H592-34987-01
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Healthy; Elderly
Keywords: healthy older people

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dried plum (Experimental): subjects will have 25% by weight (~ 600 kcal if eat 2500 kcal diet) of their usual diet substituted by dried plum powder
  Interventions: Dietary Supplement: dried plum powder

INTERVENTIONS:
Dietary Supplement: dried plum powder — subjects will have 25% of their diet substituted by dried plum powder

SUMMARY:
Dried plums (Prunus domestica L.) have traditionally been recognized for their health benefits related to conditions such as constipation, irregular menstrual cycles and mouth sores. This dried fruit provides high levels of fiber, vitamins and minerals. Dried plum has also been shown in animal studies to have beneficial effects on bone and can prevent the loss of bone caused by low hormone levels such as occurs after surgical removal of the ovaries. We also have shown that dried plum can prevent the loss of bone associated with aging in mice. Very few therapies for osteoporosis actually reverse bone loss and improve bone strength. The potential therapeutic value of dried plum in men and women with hormone deficiency or age-related osteoporosis is clear.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 yrs and 75 yrs
* Nonsmokers
* Normal renal and hepatic function

Exclusion Criteria:

* Subjects who must follow a specific diet
* Subjects on any daily medications that affect bone health
* Subjects too heavy for the DEXA machine (weight limit 300 lbs)
* Subjects whose BMD by DEXA indicates osteoporosis
* Subjects unwilling to follow the diet specified
* Pregnant women
* Subjects who are unable to understand the consent form.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
urinary calcium excretion | one month

SECONDARY OUTCOMES:
ability to tolerate the diet | one month

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Halloran, MD, Principal Investigator — SFVAMC
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Deyhim F, Stoecker BJ, Brusewitz GH, Devareddy L, Arjmandi BH. Dried plum reverses bone loss in an osteopenic rat model of osteoporosis. Menopause. 2005 Nov-Dec;12(6):755-62. doi: 10.1097/01.gme.0000185486.55758.5b. Epub 2005 Nov 8. PMID 16278620